CLINICAL TRIAL: NCT06195397
Title: Determining the Effects of an Evidence-Based Practice Education Intervention Program Applied to Nursing Students: A Randomized Controlled Trial
Brief Title: Determining the Effects of an Evidence-Based Practice Education Intervention Program Applied to Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Fatma Taş Arslan, Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SelcukU-12b-2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Evidence-Based Practice
Keywords: Evidence; Nursing Student; Evidence-Based Education

STUDY DESIGN:
Intervention Model Description: parallel group (experimental-control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): A total of 12 hours of Evidence-Based Education intervention was applied to students in the intervention group, spread over 7 sessions.
  Interventions: Other: Evidence-Based Education intervention
- No Intervention: Control Group (No Intervention): No training was given.

INTERVENTIONS:
Other: Evidence-Based Education intervention — A total of 12 hours of Evidence-Based Education intervention was applied to students in the intervention group, spread over 7 sessions.
  Arms: Experimental: Intervention Group

SUMMARY:
It was planned to evaluate the effectiveness of the evidence-based practice education intervention program in 3rd year students of the Faculty of Nursing on their knowledge, attitude, behavior and future use of evidence-based practice, and their awareness and attitudes towards research and developments.

The study was parallel group (experimental-control), randomized controlled experimental design with pretest-posttest design.

It was carried out in 3rd year students of nursing department of Selçuk University Faculty of Nursing in Konya province.

Study data were collected from 108 students between February 2023 and June 2023. Nursing students in the intervention (n = 54) and control groups (n = 54) were determined by randomization method.

DETAILED DESCRIPTION:
A total of 12 hours of Evidence-Based Education intervention was applied to students in the intervention group, spread over 7 sessions. The educational intervention was created in line with the literature. No application was given to the students in the control group. Data were collected using the Students' Knowledge, Attitudes and Behavior Towards Evidence-Based Nursing Scale and the Nursing Students' Awareness and Attitudes Towards Research and Developments in Nursing Scale.

Paired Sample T test and Wilcoxon test will be used in pre-test and post-test comparisons. Mann Whitney U, Kruskal Wallis, One Way Anova test will be applied to determine the difference between groups. Statistical significance level was accepted as p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

* Be registered in the third year of nursing
* Having taken a research course

Exclusion Criteria:

* The student suspends his/her registration or transfers to another university
* Not volunteering to participate in the study

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Knowledge, Attitude and Behavior Scale on Evidence-Based Nursing | Change from baseline and post test (after 14 weeks).
  Knowledge, Attitude and Behavior Scale on Evidence-Based Nursing The Likert-type scale consists of four sub-dimensions: "knowledge", "attitude", "future use" and "application" and 26 items. Although the scale does not have a total score, each sub-dimension is evaluated separately. A high score indicates that the student has more knowledge.
Nursing Students' Awareness and Attitude Scale to Research and Developments | Change from baseline and post test (after 14 weeks).
  The scale is a five-point Likert type (strongly disagree = 1, strongly agree = 5) and consists of 29 items, 17 of which are positive and 12 of which are negative, and has a single sub-dimensional. The scores that can be obtained from the scale vary between 29-145. A high average score indicates that awareness and positive attitude towards research is high.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Taş Arslan, PhD, Principal Investigator — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcuk University, Konya, Selcuklu
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No